CLINICAL TRIAL: NCT00888290
Title: Sodium Bicarbonate Supplementation in Chronic Kidney Disease Evaluation of Dose Response, Safety and Beneficial Effects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Michal L. Melamed, Assistant Professor, Albert Einstein College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-376
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Disease
Keywords: metabolic acidosis; chronic kidney disease; Estimated GFR 15-45
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Bicarbonate (Active Comparator): Sequential design. Participants will be getting different doses of sodium bicarbonate during the study.
  Interventions: Drug: Sodium bicarbonate
- Placebos (Placebo Comparator): Sequential design. Participants will be getting either placebo of different doses during the study.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate at 3 different doses or placebo. The different doses tested will be: 0.3 mEq/kg of ideal body weight, 0.6 mEq/kg of ideal body weight and 1 mEq/kg pf ideal body weight
  Other Names: sodium hydrogen carbonate
  Arms: Sodium Bicarbonate
Drug: Placebos — Placebo at 3 different doses to match Sodium bicarbonate dosing
  Other Names: identical-appearing placebo
  Arms: Placebos

SUMMARY:
This study will enroll 25 patients with kidney disease to evaluate the effects of different doses of sodium bicarbonate (baking soda) on levels of bicarbonate in the blood, kidney function and muscle strength. The investigators will also evaluate safety and tolerability of different doses.

DETAILED DESCRIPTION:
This study enrolled 20 patient to evaluate the effects of different doses of sodium bicarbonate. We will test serum bicarbonate levels, potassium levels and muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Estimated GFR < 45 ml/min/1.73m2 and >15 ml/min/1.73 m2 determined by abbreviated 4 variable modification MDRD equation
* Age >21

Exclusion Criteria:

* Previous chronic treatment with alkali (including sodium bicarbonate, calcium carbonate or baking soda)
* Bicarbonate level <20 or >25 mEq/L
* Decompensated heart failure
* Systolic blood pressure >160 mm/Hg
* Moderate or greater lower extremity edema
* Initiation of ESRD treatment planned within 6 months
* Kidney transplantation
* Treatment with immunosuppressives within the last 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hostetter, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine/ Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Melamed ML, Hostetter TH, Bauer C, Raff AC, Almudevar AL, Lalonde A, Messing S, Abramowitz MK. Effect of oral sodium bicarbonate on fibroblast growth factor-23 in patients with chronic kidney disease: a pilot study. BMC Nephrol. 2016 Aug 5;17(1):114. doi: 10.1186/s12882-016-0331-6. PMID 27495287
- [Result] Abramowitz MK, Melamed ML, Bauer C, Raff AC, Hostetter TH. Effects of oral sodium bicarbonate in patients with CKD. Clin J Am Soc Nephrol. 2013 May;8(5):714-20. doi: 10.2215/CJN.08340812. Epub 2013 Feb 7. PMID 23393105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will receive both active treatment and placebo. Therefore the 20 patients who started placebo also started active treatment. There are only 20 participants total in the study.
Groups:
- All Participants: Sequential design. Participants all began with taking placebo for 2 weeks and started sodium bicarbonate using escalating doses of sodium bicarbonate with a dose increase every 2 weeks (0.3 mEq/kg of ideal body weight, 0.6 mEq/kg of ideal body weight and 1 mEq/kg pf ideal body weight).
Period: Overall Study
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants went through sequential dosing of placebo, then sodium bicarbonate escalating doses.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Black | 11
  Race/ethnicity: Hispanic | 9
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 134 (13)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 70 (7)
Serum Bicarbonate Levels [Mean (Standard Deviation); unit: mEq/L] | 23.0 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Serum Bicarbonate Levels
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Sodium Bicarbonate: Crossover design. Participants will be getting different doses of sodium bicarbonate during the study.
  Sodium bicarbonate: Sodium bicarbonate at 3 different doses or placebo. The different doses tested will be: 0.3 mEq/kg of ideal body weight, 0.6 mEq/kg of ideal body weight and 1 mEq/kg pf ideal body weight
- Placebos: Crossover design. Participants will be getting either placebo of different doses during the study.
  Placebos: Placebo at 3 different doses to match Sodium bicarbonate dosing
Arm/Group | Sodium Bicarbonate | Placebos
Number analyzed (Participants) | 20 | 20
mEq/L | 25.5 (2.3) | 22.2 (2.8)

2. Secondary Outcome: Muscle Strength as Measured by sit-to Stand Test
Description: 10 repetition sit-to-stand test
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Sodium Bicarbonate | Placebos
Number analyzed (Participants) | 20 | 20
Seconds | 22.2 (1.6) | 23.8 (1.4)

3. Secondary Outcome: Systolic Blood Pressure
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Sodium Bicarbonate | Placebos
Number analyzed (Participants) | 20 | 20
mmHg | 127 [121 to 133] | 129 [122 to 139]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Sodium Bicarbonate | Placebos
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Bicarbonate (N=20) | Placebos (N=20)
Shortness of breath (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes